CLINICAL TRIAL: NCT06875453
Title: The Effect of De-tethering Exercises on Muscle Tone in Patients with Adolescent Idiopathic Scoliosis
Brief Title: De Tethering Exercises for Scolisis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burçin Akçay (Other)
Responsible Party: Sponsor-Investigator, Burçin Akçay, Associate professor, Bandırma Onyedi Eylül University
Organization: Bandırma Onyedi Eylül University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: De tethering exercises
Record Dates: First submitted 2025-03-09; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Scoliosis Idiopathic; Exercise; Muscle Tone
Keywords: scoliosis; exercise; muscle tone
MeSH Terms: conditions — Motor Activity; Scoliosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Detethering exercises will be performed for participants with adolescent idiopathic scoliosis.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The Schroth Best Practice program, which is widely used in the conservative treatment of scoliosis, consists of 6 modules including physiological exercises to correct the sagittal plane, activities of daily living, 3D correction techniques, powerful Schroth exercises, de-tethering exercises and gait rehabilitation. Detethering exercises in this program will be performed in this study.

SUMMARY:
This study aimed to investigate the effect of Detethering exercises on muscle tone in patients with adolescent idiopathic scoliosis.

H1: Detethering exercises affect muscle tone in patients with adolescent idiopathic scoliosis.

DETAILED DESCRIPTION:
This study is planned to include 15 patients diagnosed with adolescent idiopathic scoliosis.

Muscle tone and trunk rotation degree will be measured before and after the application of detethering exercises.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 10-30,
* Being diagnosed with IS
* Cobb angle between 20º and 50º,
* To be able to continue the program to be implemented,
* No chronic disease requiring the use of any neurological or psychiatric medication,
* Parents and/or child volunteering to participate in the study.

Exclusion Criteria:

* The patient has any contra-indication for exercise,
* Previous spine surgery,
* Having a curve with an apex thoracic 6 and above,
* The presence of any mental problem,
* Scoliosis is not idiopathic but has different causes (neurological, congenital, etc...), neurological, psychiatric, muscular, rheumatic or orthopedic diseases are present.

Ages: 10 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
ATR - Angle of Trunk Rotation | 1 week
  Measurement of the angle/degree of trunk rotation is the most appropriate method for the clinical evaluation of scoliosis. ATR can be used to monitor the effects of treatment without radiographic evaluation. ATR is measured using a special inclinometer called a scoliometer. The patient is asked to lean forward with arms relaxed. The scoliometer is placed on the back and the degree observed at each point of maximum gibbosity is recorded.
Muscle Tone | 1 week
  Intramuscular mechanical properties can be measured with the MyotonPRO device (Myoton Ltd., Estonia), a new diagnostic evaluation method, which measures intramuscular tension or resting muscle tone, muscle compliance, and muscle elasticity. In this study, it was shown that in conditions where electromyographic measurements are not possible, MyotonPRO measurements (viscoelastic and biomechanical properties) are used as an alternative to muscle strength and activation. The device is held upright and downward pressure is applied. When the red light on the plexiglass frame of the device probe turns green, the pressure application is stopped and the device is held stationary until 5 strokes are performed. Standard stroke intervals are used in all evaluations. During the application, care is taken to move the device and maintain the correct position. Measurements will be repeated 3 times and averaged.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandırma Onyedi Eylül University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation,, Bandırma, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No